CLINICAL TRIAL: NCT04759508
Title: " Effects of Flaxseed in Blood Pressure of Patients Taking Anti Hypertensive Drugs- A Double Blinded Placebo Controlled Randomized Trial."
Brief Title: Flaxseed in Controlling Blood Pressure of Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Rakesh Verma, Principal Investigator, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRC/1955/020
Record Dates: First submitted 2021-02-09; First posted 2021-02-18 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 500 mg BD Flax Oil Capsule with Antihypertensive drug (Active Comparator): Flax Oil Capsule 500 mg twice a day will be administered alongside antihypertensive drug in newly diagnosed hypertensive subjects
  Interventions: Dietary Supplement: Flax Oil Capsule
- Placebo(Soya Oil) Capsule with Antihypertensive drug (Placebo Comparator): No flax oil capsule,only placebo(soya oil) capsule will be administered alongside equivalent antihypertensive drug in newly diagnosed hypertensive subjects.
  Interventions: Dietary Supplement: Placebo Soya Oil Capsule

INTERVENTIONS:
Dietary Supplement: Flax Oil Capsule — Flaxseed with brand name Flax Oil Capsule will be administered to subjects receiving antihypertensives.
  Arms: 500 mg BD Flax Oil Capsule with Antihypertensive drug
Dietary Supplement: Placebo Soya Oil Capsule — Placebo capsule filled with soya oil and inert(inactive) substances will be administered to subjects remaining anti hypertensives.
  Arms: Placebo(Soya Oil) Capsule with Antihypertensive drug

SUMMARY:
Hypertension is one of the major risk factor for global mortality. Approximately half of 17 million cardiovascular deaths worldwide are accounted for HTN. Multiple research for cost-effective medication for management of hypertension is going on. An effective alternative to medications in managing hypertension is through lifestyle modifications. Adopting healthy diet is a valuable strategy. Randomized controlled year-long trials observed impressive reductions in blood pressure in patients with hypertension consuming flaxseed daily. Therefore, attention has been garnered for flaxseed as a potentially valuable strategy for the management of hypertension. Double blinded, 2 parallel-group, prospective interventional randomized clinical trial. Investigators are planning to conduct most common and basic method of randomization i.e,"lottery method". This is most popular method and simplest method. In this method both Interventional and Placebo groups are numbered on separate slips of paper of same size, shape and color. They are folded and mixed up in a drum or a box or a container. A blindfold selection is made. Required numbers of slips are selected for the desired sample size. The selection of items thus depends on chance. The respective groups are then allocated in a sequence as Code A and Code B that will be concealed from the researcher (JR) enrolling and assessing participants in sequentially numbered, opaque, sealed and stapled envelope. After getting clearance from IRC, randomization will be done where Interventional and placebo groups will be given Flaxseed Capsule 500 mg and Look-alike(Placebo) Capsule with no therapeutic effect respectively twice a day along with equivalent anti-hypertensive drugs in Medicine OPD,BPKIHS. Blood pressure of all the enrolled subjects will be taken on first day of enrollment before start of intervention. After which subjects will be given respective capsules for first 30 days then follow-up. Assigned with respective arms,subjects will be followed up on 90th day. The proforma which includes patient's sociodemographic data,BP value,Adverse Drug reactions and drug interactions will be filled and data will be entered in MS-Excel subsequently and SPSS v11.5 will be used for further analysis. Investigators are planning to conduct a clinical trial in between 2 groups using power and sample size programme. Investigators need to enroll 36 subjects in each group, to be able to reject null hypothesis that means of two different groups are equal with probability of power 95% and at 5% level of significance. Hence sample size is taken 36 in each group. 10% increment will be done in each group if the subject will not come for follow up. Clinically diagnosed hypertension attending medicine OPD, BPKIHS, Dharan, satisfying the inclusion and exclusion criteria and willing to participate in the study will be enrolled. Prior to the conduction of the study ,ethical clearance will be obtained from the Institutional Review Committee(IRC) of BPKIHS and the clinical trial will be registered. Precaution will also be taken as far as possible to avoid pain and suffering and side effects of the medication to the subjects during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age of the patient above 18 years.
2. Patients who agree to take only physician advised medicine.
3. Patient who strictly follow diet as advised.
4. Patients taking single antihypertensive drug with equivalent doses.

Exclusion Criteria:

1. Patient suffering from serious or recurrent infections.
2. Pregnancy or breast feeding women, immunodeficiency or HIV patient.
3. Patient with finding of any mental abnormality, which would interfere with or be affected by the study procedure .
4. Patient with history of bleeding disorders.
5. Hypersensitivity reaction or allergy to flaxseed.
6. History of surgery within past 6 weeks
7. Patient who do not will to give informed consent.
8. Alcohol consumption > 30 U/day..
9. Cigarette smoking > 2 pack/day
10. Patients taking multiple antihypertensive drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Flaxseed and Blood Pressure | 3 months
  Assessing the effects of Flaxseeds in systolic and diastolic blood pressure of patients taking antihypertensive drugs

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Verma, MBBS, MD, Principal Investigator — B.P. Koirala Institute of Health Sciences

IPD SHARING:
Plan to Share IPD: Yes
Individuals enrolled in the respective arms will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting February 15,2021
Access Criteria: Assess granted to sponsor, study team and data steward

REFERENCES:
- [Background] Rodriguez-Leyva D, Weighell W, Edel AL, LaVallee R, Dibrov E, Pinneker R, Maddaford TG, Ramjiawan B, Aliani M, Guzman R, Pierce GN. Potent antihypertensive action of dietary flaxseed in hypertensive patients. Hypertension. 2013 Dec;62(6):1081-9. doi: 10.1161/HYPERTENSIONAHA.113.02094. Epub 2013 Oct 14. PMID 24126178